CLINICAL TRIAL: NCT00812045
Title: A Randomised, Double-Blind, Placebo-Controlled, Parallel Group, Phase II Study to Assess the Efficacy of 28 Day Oral Administration of AZD1236 in Adult Patients With Cystic Fibrosis
Brief Title: Study to Assess Efficacy of AZD1236 in Patients With Cystic Fibrosis
Acronym: CYBER
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Andrew J Lockton, MD, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D4260C00008
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Cystic Fibrosis
Keywords: Induced sputum; cystic fibrosis; biomarker; CYBER
MeSH Terms: conditions — Cystic Fibrosis | interventions — 4-((5-chloro-2-pyridinyl)oxy)-1-((((4S)-4-methyl-2,5-dioxo-4-imidazolidinyl)methyl)sulfonyl)-piperidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD1236
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1236 — Oral tablet, 75 mg twice daily during 4 weeks
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effect of AZD1236 in patients with cystic fibrosis (CF) on inflammatory biomarkers in induced sputum, after a treatment period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Have a clinical diagnosis of cystic fibrosis with an FEV1 >40% of predicted normal
* Be able to comply with induced sputum procedure
* post-menopausal surgically sterile female (total hysterectomy and /or bilateral total oophorectomy)

Exclusion Criteria:

* Concomitant diagnosis of significant pulmonary disease other than CF-related lung disease, including symptomatic asthma and allergic bronchopulmonary aspergillosis
* Treatment with any immunomodulatory agents within 8 weeks prior to Visit 2
* Known to be infected with Burkholderia cepacia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2009-12; Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Effect on biomarker levels in induced sputum | 2 times at baseline and after 4 weeks treatment
Signs and symptoms (Lung function variables by spirometry, symptom scores from Diary and Health-related quality of life Questionnaire) | At inclusion, at randomisation and after 4 weeks treatment

SECONDARY OUTCOMES:
Safety and tolerability (adverse events, vital signs and laboratory safety variables) | throughout study (at inclusion, randomisation, after 4 weeks treatments and at follow-up)
Effect on biomarkers in blood | 2 times, at baseline and after 4 weeks treatment
Effect on biomarkers in urine | 2 times, at baseline and after 4 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Lockton, MD, Study Director — AstraZeneca R&D Charnwood; Shawn Aaron, MD, Principal Investigator — The Ottawa Hospital
Locations (10):
- Canada (3):
  - Research Site, Montreal
  - Research Site, Ottawa
  - Research Site, Vancouver
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Utrecht
- Poland (2):
  - Research Site, Gdansk
  - Research Site, Poznan
- Spain (2):
  - Research Site, Barcelona, Catalonia
  - Research Site, Madrid, Madrid